CLINICAL TRIAL: NCT03404375
Title: Validating a New Method to Assess Estimated Blood Loss in the Obstetric Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-0248
Record Dates: First submitted 2017-12-08; First posted 2018-01-19 (Actual); Results first posted 2021-02-25 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-01

CONDITIONS: Pregnancy Complications
Keywords: scheduled cesarean section; term pregnancy; estimated blood loss; postpartum hemorrhage
MeSH Terms: conditions — Pregnancy Complications; Postpartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Term patients (Other): This study only has one arm: term pregnant patients scheduled for cesarean sections. The surgeon will clinically estimate blood loss and the research team will estimate blood loss using the Gauss Triton system. This will be done on all 242 patients.
  Interventions: Device: Gauss Triton system

INTERVENTIONS:
Device: Gauss Triton system — The Triton system (Gauss Surgical, Inc., Palo Alto, CA) is a novel mobile monitoring platform that combines mobile computing with Gauss Feature Extraction Technology (FET) to directly assess Hb mass (mHb) absorbed by surgical sponges from an image. The device is an iPad like imaging device that will assess blood loss via imaging of the surgical sponges used in the surgery.
  The device will be used to calculate blood loss on every patient enrolled in the study.

SUMMARY:
Postpartum hemorrhage (PPH) is the leading cause of maternal mortality in low-income countries and the primary cause of nearly one quarter of all maternal deaths globally. Estimates of blood loss at delivery are notoriously inaccurate, with under-estimation more common than over-estimation. Traditionally, the surgeon performing the cesarean section would estimate the blood loss by visually assessing the blood collected in the surgical drape and counting the number of lap sponges used thru out the procedure. The investigators would like to study and validate an FDA approved device called the gauss Triton device used to estimate blood loss during scheduled cesarean sections.

DETAILED DESCRIPTION:
According to the World Health Organization, postpartum hemorrhage (PPH) is the leading cause of maternal mortality in low-income countries and the primary cause of nearly one quarter of all maternal deaths globally. An estimated blood loss (EBL) in excess of 500 mL following a vaginal birth or a loss of greater than 1,000 mL following cesarean birth often have been used for the definition of postpartum hemorrhage, but the average volume of blood lost at delivery can approach these amounts when actually measured rather than estimated. More than half of all maternal deaths occur within 24 hours of delivery, most commonly from excessive bleeding. Worldwide, 140,000 women succumb to postpartum hemorrhage each year. The most common antecedents to postpartum hemorrhage are uterine atony, placental disorders, and trauma during delivery. Improving maternal health worldwide is one of the WHO's 8 Millennium Developmental Goals. The prevention and treatment of PPH is an essential step towards the achievement of that goal.

Estimates of blood loss at delivery are notoriously inaccurate, with under-estimation more common than over-estimation. Traditionally, the surgeon performing the cesarean section would estimate the blood loss by visually assessing the blood collected in the surgical drape and counting the number of lap sponges used thru out the procedure. Current detection and management of hemorrhage is heavily based on clinical judgment, which often leads to delay in recognition and intervention. Often, interventions such as fluid resuscitation and blood transfusion are not initiated until significant hemorrhage has already taken place. The traditional method for estimating blood loss is based on the surgeon and surgical staff's subjective assessment that is severely limited by human error and the presence of large volumes of amniotic fluid, irrigation, or both. Another limitation is that blood loss is frequently estimated at the end of the procedure.

Early detection and treatment of this potentially life threatening obstetric complication is of utmost importance in the field of obstetrics. Simulations and didactic training have been shown to improve visual estimations, but there are still poor associations between experience level and accuracy, and a significant decay in blood loss estimation skills over time.

The Triton system (Gauss Surgical, Inc., Palo Alto, CA) is a novel mobile monitoring platform that combines mobile computing with Gauss Feature Extraction Technology (FET) to directly assess Hb mass (mHb) absorbed by surgical sponges from an image. The device is an iPad like imaging device that will assess blood loss via imaging of the surgical sponges used in the surgery. In 2014, Konig at al. showed that mobile blood loss monitoring using the Triton system is accurate in assessing mHb on surgical sponges across a range of ambient light conditions, sponge saturation, saline contamination, and initial blood Hb. Utilization of this tool could significantly improve the accuracy of blood loss estimates. Holmes et al. also showed that the novel mobile monitoring system provides an accurate measurement of mHb on surgical sponges as compared with manual rinsing measurements, and is significantly more accurate than the gravimetric method.

However, these studies were performed on patients undergoing a myriad of surgical procedures not just limited to obstetrical patients. To the investigators' knowledge, this technology has not been validated in the obstetrical population at risk for hemorrhage.

The gauss/triton colorimetric system is not standard of care at UTMB. Not enough data is available to support its use, despite being FDA approved to estimate blood loss. Most evidence is available in non-pregnant patients. In the obstetric population no definitive evidence exists, and the only trial that has been performed was recently published in AJP reports. In that trial, only the accuracy was evaluated, and the investigators believe that further evidence is needed to support its use.

The investigators' hypothesis is that this device will enable clinicians to prospectively and objectively assess EBL. Ultimately after its validation, their results will be used to propose a multicenter clinical trial to the NICHD MFMU network to evaluate the clinical utility of this system.

This study will be a prospective cohort study, in which the investigators will evaluate two methods of evaluating intraoperative blood loss during cesarean delivery (usual clinical assessment versus Device). Of note, the subjects consented will be used as self-controls. Patients who are scheduled for an elective cesarean and meet criteria for inclusion in the study will be approached for participation at same day of admission. Written informed consent will be obtained from the patients. If patients agree to participate, a CBC (complete blood count) will be obtained via venous puncture. The device will be used during the delivery in the operating room. The device will be used to assess EBL by the research staff only and results/ EBL assessment will be masked to the clinical team. Unmasking will only occur after collecting the data from the device with purpose to perform data analysis. Patient management will be according to the clinical team. All patients undergo a CBC postpartum. The drop in Hgb (ΔHgb) between the pre and post cesarean CBCs will be calculated for each patient. Patients will be divided into quartiles of ΔHgb. Cases will be those patients whose ΔHgb is in the upper quartile, while controls will be those patients whose ΔHgb is in the lower 3 quartiles. The investigators will be comparing EBL by standard clinical assessment versus result from the device between cases and controls.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between the ages of 18-50
* Scheduled cesarean delivery

Exclusion Criteria:

* Incarcerated patients
* Patient unwilling or unable to provide consent
* Intrauterine fetal demise (no fetal heart beat identified and documented by two physicians)
* Placenta previa or other known placental anomalies
* Enrolled in another trial that may affect outcome.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Term pregnant patients scheduled for cesarean section
Enrollment: 242 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fawzi Saoud, MD, Principal Investigator — UTMB-Galveston
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Saoud F, Stone A, Nutter A, Hankins GD, Saade GR, Saad AF. Validation of a new method to assess estimated blood loss in the obstetric population undergoing cesarean delivery. Am J Obstet Gynecol. 2019 Sep;221(3):267.e1-267.e6. doi: 10.1016/j.ajog.2019.06.022. Epub 2019 Jun 20. PMID 31229429

RESULTS

PARTICIPANT FLOW:
Groups:
- Cases: Cases defined as delta hemoglobin in the upper quartile
- Control: Controls defined as delta hemoglobin in the lower quartile
Period: Overall Study
Arm/Group | Cases | Control
Started | 70 | 172
Completed | 70 | 172
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cases | Control | Total
Number analyzed (Participants) | 70 | 172 | 242
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 30 [27 to 35] | 29 [25 to 34] | 29 [25 to 35]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 172 | 242
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 69 | 95
  Not Hispanic or Latino | 44 | 103 | 147
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 70 | 172 | 242

OUTCOME MEASURES:

1. Primary Outcome: Clinical Estimated Blood Loss (EBL) Between Cases and Controls Using Clinical Estimate Versus Device Assessment
Description: The investigators are looking at the difference between the EBL measured clinically and the EBL measured using the Gauss device
Time Frame: 48 hours
Measure: Median (Inter-Quartile Range); unit: milliLiters
Arm/Group | Cases | Control
Number analyzed (Participants) | 70 | 172
milliLiters | 800 [700 to 900] | 800 [600 to 900]

2. Secondary Outcome: Transfusion Requirements
Description: Number of participants that received blood transfusion
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Cases | Control
Number analyzed (Participants) | 70 | 172
Participants | 0 | 1

3. Secondary Outcome: Number of Participants With Post-partum Hemorrhage
Description: the number of cases of post partum hemorrhage
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Cases | Control
Number analyzed (Participants) | 70 | 172
Participants | 8 | 11

4. Primary Outcome: Triton Device Estimated Blood Loss (EBL) Between Cases and Controls Using Clinical Estimate Versus Device Assessment
Description: The investigators are looking at the difference between the EBL measured clinically and the EBL measured using the Gauss device (Triton)
Time Frame: 48 hours
Measure: Median (Inter-Quartile Range); unit: milliLiters
Arm/Group | Cases | Control
Number analyzed (Participants) | 70 | 172
milliLiters | 474 [300 to 642] | 331 [222 to 469]

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Cases | Control
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/172
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/172
Other Adverse Events (participants affected / at risk) | 8/70 | 11/172
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cases (N=70) | Control (N=172)
Post Partum Hemorrhage (Blood and lymphatic system disorders) | 8 (8) | 11 (11) — Number of participants with blood loss of > 1000 mL

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/75/NCT03404375/Prot_SAP_000.pdf